CLINICAL TRIAL: NCT01832740
Title: Impact of Transcranial Slow Oscillating Stimulation on Memory Consolidation During Nocturnal Slow Wave Sleep in Younger, Healthy Subjects
Brief Title: Effects of Brain Stimulation During Nocturnal Sleep on Memory Consolidation in Younger, Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Agnes Flöel, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Nighttime sleep-tSOS-Young
Record Dates: First submitted 2013-03-08; First posted 2013-04-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Subjects
Keywords: young healthy subjects; brain stimulation; tSOS; tDCS; sleep; memory; memory consolidation
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0,75 Hz stimulation (Experimental): slow transcranial oscillating stimulation (~0,75Hz) during periods of Slow Wave Sleep
  Interventions: Device: brain stimulation
- SHAM stimulation (Experimental): SHAM stimulation during periods of Slow Wave Sleep
  Interventions: Device: SHAM

INTERVENTIONS:
Device: brain stimulation — oscillating direct current brain stimulation
  Arms: 0,75 Hz stimulation
Device: SHAM — no stimulation
  Arms: SHAM stimulation

SUMMARY:
The beneficial effect of nocturnal sleep on memory consolidation is well-documented in young, healthy subjects. Especially, periods rich in slow-wave sleep (SWS) have shown a memory enhancing effect on hippocampus-dependent declarative memory. Slow oscillatory activity typically occuring during SWS has been implicated in the consolidation effect. In this study we investigate if the consolidation effect can be amplified by the application of a weak transcranial oscillatory electric current within the frequency range of SWS in humans (0,7-0,8 Hz) during nocturnal SWS.

ELIGIBILITY:
Inclusion Criteria:

* healthy Subjects
* unobtrusive, neuropsychological screening
* age: 18-35 years
* right handed

Exclusion Criteria:

* untreated severe internal or psychiatric diseases
* epilepsy
* other severe neurological diseases eg., previous major stroke, brain tumour
* contraindications to MRI

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Retention of declarative memories after 0.75 Hz stimulation during SWS, vs after sham stimulation during SWS | 4 weeks
  Retention (difference values between performance at retrieval after sleep minus performance at learning before sleep) between stimulation conditions (0.75 Hz during SWS, vs sham stimulation during SWS) in the declarative memory task.

SECONDARY OUTCOMES:
1. Amount of Slow wave Sleep | 4 weeks
  1. Amount of slow wave sleep assessed by standard polysomnographic criteria in 0,75 Hz vs SHAM stimulation during SWS.
2. sleep spindels | 4 weeks
  2. Spindel activity during sleep indicated via several spindel parameters like number, duration, frequency of spindles; compared between 0,75 Hz and SHAM stimulation during SWS.
3. EEG-correlates | 4 weeks
  3. Neuronal correlates (EEG-power in slow oscillation frequency bands induced by 0,75 Hz vs SHAM stimulation during SWS; EEG-correlates of encoding and retrieval of a declarative memory task).
4. further memory systems | 4 weeks
  4. Performance in further memory systems (procedural), compared between 0,75 Hz and SHAM stimulation during SWS.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Professor, Principal Investigator — Charite Universitätsmedizin Berlin - Neurologie
Locations (1):
- Charite CCM Neurologie Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Marshall L, Helgadottir H, Molle M, Born J. Boosting slow oscillations during sleep potentiates memory. Nature. 2006 Nov 30;444(7119):610-3. doi: 10.1038/nature05278. Epub 2006 Nov 5. PMID 17086200
- [Background] Diekelmann S, Born J. The memory function of sleep. Nat Rev Neurosci. 2010 Feb;11(2):114-26. doi: 10.1038/nrn2762. Epub 2010 Jan 4. PMID 20046194